CLINICAL TRIAL: NCT06746805
Title: The Effect of Acute Ketone Monoester Supplementation on Glucose Oxidation During Exercise Performed With High Rates of Carbohydrate Ingestion in Trained Cyclists
Brief Title: The Effect of Acute Ketone Monoester Supplementation on Glucose Oxidation During Exercise
Acronym: KETONE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: METC 23-001
Record Dates: First submitted 2024-03-11; First posted 2024-12-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-05

CONDITIONS: Exercise Metabolism

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled, cross-over trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Color and flavor matched placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CHO+KETONE (Experimental): Interventional drink with glucose + ketone monoester
  Interventions: Dietary Supplement: CHO+KETONE
- CHO+PLACEBO (Placebo Comparator): Placebo drink with glucose + placebo
  Interventions: Dietary Supplement: CHO+PLACEBO

INTERVENTIONS:
Dietary Supplement: CHO+KETONE — Sports drink containing glucose and ketone mono-esters
  Arms: CHO+KETONE
Dietary Supplement: CHO+PLACEBO — Sports drink containing glucose and placebo
  Arms: CHO+PLACEBO

SUMMARY:
The purpose of this study is to examine the effect of exogenous ketone body supplementation on carbohydrate metabolism during exercise. In a randomized, crossover, and double-blind study, 20 endurance trained adult males and females aged 18-50 years, will ingest carbohydrates with either a ketone monoester supplement before and throughout a 3-hour exercise session or carbohydrates with a flavour-matched ketone-free placebo. The main aim of this study is to compare the exogenous carbohydrate oxidation rates during exercise between the ketone monoester and placebo conditions.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Trained cyclist/triathlete (VO2peak > 55 ml/kg/min for males and >48 ml/mg/min for females)
* Healthy as per medical history and investigator's/physician's judgement
* Having given written informed consent

Exclusion Criteria:

* Use of medication that could impact study outcomes and/or interfere with the expected mechanism of action of ketone supplements (e.g. Chronic use of gastric acid suppressing medication, statins, corticosteroids)
* Smoking
* Diagnosed acute or chronic medical conditions that, in the opinion of the investigator, could impact study outcomes (e.g. Diabetes mellitus)
* Diagnosed musculoskeletal disorders
* Adhering to a carbohydrate restrictive diet
* Participation in another study at the same time
* Blood donation in the 2 months before the first experimental trial
* Plasma donation in the 2 weeks before the first experimental trial
* Males: VO2peak <55 ml/min/kg body mass
* Females: VO2peak <48 ml/min/kg body mass
* Females: pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Exogenous carbohydrate oxidation rate | Acute:during 3 hours of exercise
  Exogenous carbohydrate oxidation rate during exercise measured by 13C enrichment in breath. CHO+KETONE vs CHO+PLACEBO condition

SECONDARY OUTCOMES:
Endogenous carbohydrate disappearance rate | Acute:during 3 hours of exercise
  Endogenous carbohydrate disappearance rate during exercise measured by stable isotope tracer methodology. CHO+KETONE vs CHO+PLACEBO condition
Exogenous carbohydrate disappearance rate | Acute:during 3 hours of exercise
  Exogenous carbohydrate disappearance rate during exercise measured by stable isotope tracer methodology. CHO+KETONE vs CHO+PLACEBO condition
Total carbohydrate disappearance rate | Acute:during 3 hours of exercise
  Total carbohydrate disappearance rate during exercise measured by stable isotope tracer methodology. CHO+KETONE vs CHO+PLACEBO condition
Exogenous carbohydrate appearance rate | Acute:during 3 hours of exercise
  Exogenous carbohydrate appearance rate during exercise measured by stable isotope tracer methodology. CHO+KETONE vs CHO+PLACEBO condition
Endogenous carbohydrate appearance rate | Acute:during 3 hours of exercise
  Endogenous carbohydrate appearance rate during exercise measured by stable isotope tracer methodology. CHO+KETONE vs CHO+PLACEBO condition
Total carbohydrate appearance rate | Acute:during 3 hours of exercise
  Total carbohydrate appearance rate during exercise measured by stable isotope tracer methodology. CHO+KETONE vs CHO+PLACEBO condition
Plasma glucose enrichments during exercise | Acute:during 3 hours of exercise
  Plasma glucose enrichments during exercise measured by stable isotope tracer methodology. CHO+KETONE vs CHO+PLACEBO condition

OTHER OUTCOMES:
Total carbohydrate oxidation | Acute:during 3 hours of exercise
  Total carbohydrate oxidation during exercise, measured indirectly by using traditional stoichiometric calculations of carbohydrate oxidation. CHO+KETONE vs CHO+PLACEBO condition
Blood parameters | Acute:during 3 hours of exercise
  Plasma glucose, insulin, glycerol, free fatty acids, and ketone body concentrations (including area under the curve) following drink ingestion. CHO+KETONE vs CHO+PLACEBO condition
Exercise economy during cycling | Acute:during 3 hours of exercise
  Exercise economy during the exercise trial. CHO+KETONE vs CHO+PLACEBO condition, will be determined based on the amount of work performed during cycling (workload), and the amount of energy expenditure as measured by indirect calorimetry.
Exercise heart rate | Acute:during 3 hours of exercise
  Heart rate during exercise. CHO+KETONE vs CHO+PLACEBO condition

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available upon request